CLINICAL TRIAL: NCT05617157
Title: Effects of Stair Stepping on Late Day Postprandial Glycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jochen Kressler, Associate Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS-2022-0184
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Glycemic Control

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Stair stepping (Experimental)
  Interventions: Other: Stair stepping

INTERVENTIONS:
Other: Stair stepping — stepping up and down 32 stairs for 1 minute
  Arms: Stair stepping

SUMMARY:
1. Purpose/objective:

   The purpose of the current study is to investigate whether the benefits of stair stepping established for early day food consumption extend to late day food consumption.
2. Methods:

   Participants will perform two standard oral glucose tolerance test (OGTT), consuming 75g of glucose dissolved in 350mL of water followed by assessment of glycemic markers for 2 hours. Participants will perform the OGTTs in the evening of two separate days. One day will be the control condition, where participants will remain seated throughout the entire duration of the OGTT. The other day (in randomized order) participants will perform 1 min of stair stepping at a self-selected, comfortable pace 28min after the consumption of the glucose solution. Blood glucose measurement via standard, over the counter finger sticks will be performed every 10 min for the first hour, and again at 90 and 120min of the OGTT. In addition, standard venipuncture blood draws (5mL) will be drawn at baseline ad at peak (30min) glucose excursion for the assessment of insulin. Participants will be instructed to not vary their diet or exercise during the two testing days. Diet and activity logs will be collected and analyzed to verify compliance.
3. Subjects Adults 18 or over will be recruited for this project. Prior to enrolling in the study, each potential participant will complete the Physical Activity Recall Questionnaire (PAR-Q+) to screen for cardiovascular risks. Any positive responses to questions from the PAR-Q+ will eliminate the individual from selection. Participants who self report any condition that will prevent them form safely and/or comfortably climbing stairs will also be excluded form participation.
4. Planned analyses: Results will be analyzed via a 2-factor repeated measure analysis of variance for time and condition. Statistical significance will be set at an alpha level of 0.05.
5. Potential benefits:

   This study will help to identify the shortest possible bout of exercise that is still effective in significantly reducing postprandial blood glucose using a simple, cheap, and ubiquitously available exercise mode - stair stepping. In addition, participants will be informed of their fasting and postprandial glycemic response if they so desire. At the end of the study, individuals that want their test results will be given a copy. However, we cannot guarantee the subjects will benefit from this information.
6. Potential risks:

Risks are comparable to regular everyday life. Stair stepping performed in this study presents the same risk of falling or errant stepping related injuries as any other stair stepping at a comfortable pace. Finger sticks and venipunctures present no greater risk than a regular routine physical examination. Whenever blood is drawn, there is a small risk of bruising or infection.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy individuals able to stair step for 1 minute

Exclusion Criteria:

* Prior to enrolling in the study, each potential participant will complete the Physical Activity Recall Questionnaire (PAR-Q+) to screen for cardiovascular risks. Any positive responses to questions from the PAR-Q+ will eliminate the individual from selection.
* Participants who self report any condition that will prevent them form safely and/or comfortably climbing stairs will also be excluded form participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose | 0-120 minutes after 75g of glucose consumption
  Plasma Glucose

SECONDARY OUTCOMES:
Insulin | 0 and 60 minutes after 75g of glucose consumption
  Insulin

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States